CLINICAL TRIAL: NCT01602302
Title: Ultrasound as Biomarker for Withdrawal of Biological DMARDs in Rheumatoid Arthritis
Brief Title: Ultrasound and Withdrawal of Biological DMARDs in Rheumatoid Arthritis
Acronym: RA-BioStop
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: low recruitment
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Dejaco Christian, MD, PD, Dr., Medical University of Graz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-5; V2; 2011-005204-15 (EudraCT Number)
Record Dates: First submitted 2012-05-16; First posted 2012-05-18 (Estimated); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; ultrasound; remission; biological DMARD
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept; Adalimumab; Infliximab; Certolizumab Pegol; golimumab; Abatacept; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm ( bDMARD withdrawal ) (Experimental): single arm (bDMARD withdrawal)
  Interventions: Drug: bDMARD withdrawal (etanercept, adalimumab, infliximab, certolizumab, golimumab, tozilizumab, abatacept)

INTERVENTIONS:
Drug: bDMARD withdrawal (etanercept, adalimumab, infliximab, certolizumab, golimumab, tozilizumab, abatacept) — bDMARDS (etanercept, adalimumab, infliximab, certolizumab, golimumab, tocilizumab, abatacept) will be discontinued after baseline visit in all participants
  Other Names: Enbrel; Humira; Remicade; Cimzia; Simponi; Roactemra; Orencia

SUMMARY:
biological DMARDs may be stopped in Rheumatoid Arthritis (RA) patients treated with a combination of synthetic DMARD plus bDMARDs which are in persistent clinical remission. The research question of this study is, whether musculoskeletal sonography is a useful biomarker predicting a disease flare after cessation of bDMARD therapy.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is the most common inflammatory joint disease. It is usually treated with synthetic and biologic disease modifying antirheumatic drugs (DMARDs). Up to 35% of patients can achieve clinical remission by the combination these therapies; however, there is considerable uncertainty regarding the management of patients once this clinical state is achieved. The discontinuation of biological agents in patients with persistent clinical remission may be beneficial for the patients and the health care system reducing the risks of long term adverse events and saving costs, respectively. Up to 60% of patients were reported to flare after cessation of anti-tumor necrosis factor alpha (TNF alpha) therapy despite continuation of synthetic DMARDs and up to now there exist no validated biomarkers that predict which patients will suffer a flare and which patients will remain in remission.

Sonography is more and more used as a biomarker in RA. Subclinical inflammation was previously associated with an increased risk for short term clinical relapse and structural deterioration.

The hypothesis of this prospective study is that ultrasound verified subclinical inflammation at the time of bDMARD withdrawal predicts a disease flare at week 16. The investigators plan to recruit RA-patients with persistent clinical remission according to SDAI and no current corticosteroid therapy. At baseline, bDMARD is stopped, synthetic DMARDs are continued. Patients undergo 9 study visits within 52 weeks. Ultrasound examinations of 14 joints as well as clinical and laboratory assessments with calculation of SDAI scores are performed at each visit. Patients are considered to have a disease flare if disease status changes from remission to active disease according to clinical scores. Patients with a flare of the disease are excluded from the active phase of the study and are treated according to current guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient ≥18 years and <90 years of age
* Classification of RA according to the ACR/EULAR 2010 criteria
* Persistent clinical remission as defined by the ACR/EULAR remission criteria for at least 6 months (documented at ≥2 visits)
* Written informed consent
* Current treatment with a single csDMARD or a combination of csDMARDs plus a stable dose and administration interval (for the last 6 months) of a TNF-alpha inhibitor
* No current systemic corticosteroid treatment (stopped for at least 4 weeks), no corticosteroid injection within 4 weeks
* Stable dose of NSAIDs for at least 1 week

Exclusion Criteria:

* • Current treatment with any investigational drug
* Current administration interval of the anti-TNF-alpha agent of >11 weeks
* Complete destruction of any joint to be investigated by sonography
* Current RA-related vasculitis or other active systemic (i.e. extraarticular) RA- manifestation with the exception of rheumatoid nodules
* Initial arthritis manifestations before the age of 17 years
* Planned surgery within the study period or history of surgery of any of the joints to be investigated clinically or by sonography
* Current severe medical illness requiring hospitalization
* Active infection or active malignancy at screening or infection during the past 4 weeks requiring (even temporary) discontinuation of the anti-TNF-alpha agent
* Pregnancy or lactation
* Inability of the patient to follow the protocol
* Current treatment with Rituximab (MabThera®)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-06; Primary Completion 2020-11-19 (Actual); Study Completion 2020-11-19 (Actual)

PRIMARY OUTCOMES:
PD-signals predict relapse at week 16 | 16 weeks
  Active inflammation at the time of bDMARD withdrawal indicated by the presence of a PD-score ≥1 in at least one joint out of a sonographic 14-joint count predicts relapse rate at week 16.

SECONDARY OUTCOMES:
PD-signals predict relapse at week 24 | 24 weeks
  Active inflammation at the time of bDMARD withdrawal indicated by the presence of a PD-score ≥1 in at least one joint out of a sonographic 14-joint count predicts relapse rate at week 24
PD-signals predict relapse at week 52 | 52 weeks
  Active inflammation at the time of bDMARD withdrawal indicated by the presence of a PD-score ≥1 in at least one joint out of a sonographic 14-joint count predicts relapse rate at week 52
PD-scores at time of relapse | 24 weeks
  RA-patients have higher PD-scores at time of a clinical flare compared to patients with maintained clinical remission
Increment of PD-scores precede flare | 52 weeks
  An increment of PD-scores at follow-up compared to baseline visits precedes a clinical flare
PD scores better predict a relapse than residual swollen joints | 16, 24, 52 weeks
  PD scores better predict a relapse at week 16, 24 and 52 than the presence of residual swollen joints
PD score at baseline correlates with relapse risk | 52 weeks
  The higher the PD score at baseline, the more likely is a relapse at weeks 16, 24 and/or 52
7. Patients converting from a rheumatoid factor (RF) positive to a RF negative status are less likely to experience a relapse at weeks 16, 24 and 52 than patients remaining seropositive | 16, 24, 52 weeks
  7. Patients converting from a rheumatoid factor (RF) positive to a RF negative status are less likely to experience a relapse at weeks 16, 24 and 52 than patients remaining seropositive
8. Blood biomarkers predict the time to flare after bDMARD withdrawal
  8. Blood biomarkers predict the time to flare after bDMARD withdrawal
9. Blood biomarkers predict the time to re-achieve remission after flare and re-induction of bDMARD treatment
  9. Blood biomarkers predict the time to re-achieve remission after flare and re-induction of bDMARD treatment
PD-scores and blood biomarkers at baseline predict radiographic progression at week 52 | 52
  PD-scores and blood biomarkers at baseline predict radiographic progression at week 52

CONTACTS AND LOCATIONS:
Overall Officials: Christian Dejaco, MD, PhD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University Graz, Graz, Austria